CLINICAL TRIAL: NCT02613039
Title: Study on the Effect of Combined Oral Contraceptive Therapy on Female Sexuality, Body Image and Mental Health
Brief Title: Oral Contraceptive Therapy and Sexuality
Acronym: COSEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Mario Maggi, Full professor of Endocrinology, University of Florence
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANDRO-AOUC-2015-2
Record Dates: First submitted 2015-11-18; First posted 2015-11-24 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Contraceptive Usage; Sexual Behavior; Mental Health Wellness 1
Keywords: oral contraceptives; female sexuality
MeSH Terms: conditions — Contraception Behavior; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- female outpatient subjects (Other): Patients requiring combined Oral Contraceptives therapy.
  Interventions: Drug: Combined Estrogen-Progestin Oral Contraceptives

INTERVENTIONS:
Drug: Combined Estrogen-Progestin Oral Contraceptives — All patients enrolled will undergo Combined Estrogen-Progestin Oral Contraceptives. Different compounds will be chosen according to the approved indications and clinical practice. Therefore it is not possible to provide a specific trade and/or generic name.

SUMMARY:
Oral contraceptives (OCs) ameliorate hyperandrogenism and regulate menstrual cycles. To reduce androgenic side effects of first- and second-generation progestins, several new progestins derived from progesterone or spironolactone have been developed in the last few decades. These progestins, such as drospirenone, cyproterone acetate and NOMAC, are designed to bind specifically to the progesterone receptor and to have no androgenic, estrogenic or glucocorticoid actions.

However, OCs with a more pronounced anti-androgenic effects are more likely to induce sexual dysfunction, mainly hypoactive sexual desire disorder, which can highly impact patient and partner's quality of life. Moreover, available data indicate that OC use might increase adiposity in adolescents and might be associated with central redistribution of body fat in young women with Polycystic ovary syndrome (PCOS) without a recognizable difference in clinical anthropometric measurements, including body mass index and waist circumference.

In this context, it would be worth to evaluate the effects of combined OCs on metabolic and sexual health (sexual desire, arousal, and other parameters of sexual health), body image and mood.

DETAILED DESCRIPTION:
Primary study objective Evaluation, in a sample of female outpatient subjects, of the effect of oral contraceptives (OCs) on sexual function and distress, evaluated with the FSFI (Female Sexual Function Index) and FSDS (Female Sexual Distress Scale Revised) questionnaires and through clitoris artery hemodynamic parameters.

Secondary study objectives

Evaluation, in a sample of female outpatient subjects, of the effect of OCs on:

* body image perception, evaluated with the BUT (Body Uneasiness Test) questionnaire;
* mood and mental status, evaluated with the MHQ (Middlesex Hospital questionnaire);
* hormonal and metabolic parameters.

Exploratory Objectives: evaluation of the relationships between hormonal parameters, clinical scores and sexual function, body image, mood in the study population.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects aged =/> 18 years and of reproductive age.
* Capacity to give consent for study participation, after being adequately informed of the aims, benefits, risks, time and motion of the study.

Exclusion Criteria:

* Participation in another clinical trial.
* Known or suspected (or history of) malignancy or chronic illness.
* Serious organic or mental disease diagnosed by a psychiatrist (e.g., major depression currently treated with antidepressant medication) suspected on the basis of the medical history and/or clinical examination.
* Conditions that may affect the compliance to the study.
* Contraindications to therapy with the study drug or hypersensitivity to the study drug (active ingredient or excipients of the formulation).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10; Primary Completion 2018-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Changes in sexual function (FSFI score) | 6 months and 12 months
  A significant difference in FSFI score evaluated at baseline compared with follow-up visits will be considered as a primary endpoint.
Changes in sexual distress (FSDS score) | 6 months and 12 months
  A significant difference in FSDS score evaluated at baseline compared with follow-up visits will be considered as a primary endpoint.
Changes in clitoris vascularization | 6 months and 12 months
  A significant difference in clitoris artery hemodynamic parameters evaluated at baseline compared with follow-up visits will be considered as a primary endpoint.

SECONDARY OUTCOMES:
Changes in body image perception | 6 months and 12 months
  A significant difference in BUT score evaluated at baseline compared with follow-up visits will be considered as a primary endpoint.
Changes in mood and mental status | 6 months and 12 months
  A significant difference in MHQ score evaluated at baseline compared with follow-up visits will be considered as a primary endpoint.
Changes in glycaemia | 6 months and 12 months
  A significant difference in glycaemia levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in glycated hemoglobin (HbA1c) levels | 6 months and 12 months
  A significant difference in HbA1c levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in insulin levels | 6 months and 12 months
  A significant difference in insulin levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in total cholesterol levels | 6 months and 12 months
  A significant difference in total cholesterol levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in HDL (high-density lipoprotein) cholesterol levels | 6 months and 12 months
  A significant difference in HDL cholesterol levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in triglycerides levels | 6 months and 12 months
  A significant difference in triglycerides levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in total testosterone levels | 6 months and 12 months
  A significant difference in total testosterone levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in estradiol levels | 6 months and 12 months
  A significant difference in estradiol levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in SHBG (sex hormone binding globulin) levels | 6 months and 12 months
  A significant difference in SHBG levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in LH (luteinizing hormone) levels | 6 months and 12 months
  A significant difference in LH levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in FSH (follicle-stimulating hormone) levels | 6 months and 12 months
  A significant difference in FSH levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in prolactin levels | 6 months and 12 months
  A significant difference in prolactin levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in delta4-androstenedione levels | 6 months and 12 months
  A significant difference in delta4-androstenedione levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.
Changes in Dehydroepiandrosterone sulfate (DHEAS) levels | 6 months and 12 months
  A significant difference in DHEAS levels evaluated at baseline visit and at follow-up visits (6 or 12 months) will be considered as a secondary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Maggi, Principal Investigator — University of Florence
Locations (1):
- Ambulatori di Medicina della Sessualità e Andrologia, Florence, Italy

REFERENCES:
- [Background] Battaglia C, Battaglia B, Mancini F, Nappi RE, Paradisi R, Venturoli S. Moderate alcohol intake, genital vascularization, and sexuality in young, healthy, eumenorrheic women. A pilot study. J Sex Med. 2011 Aug;8(8):2334-43. doi: 10.1111/j.1743-6109.2011.02310.x. Epub 2011 May 19. PMID 21595833
- [Background] Battaglia C, Nappi RE, Mancini F, Cianciosi A, Persico N, Busacchi P, Facchinetti F, de Aloysio D. Menstrual cycle-related morphometric and vascular modifications of the clitoris. J Sex Med. 2008 Dec;5(12):2853-61. doi: 10.1111/j.1743-6109.2008.00972.x. Epub 2008 Aug 28. PMID 18761595
- [Background] Bullivant SB, Sellergren SA, Stern K, Spencer NA, Jacob S, Mennella JA, McClintock MK. Women's sexual experience during the menstrual cycle: identification of the sexual phase by noninvasive measurement of luteinizing hormone. J Sex Res. 2004 Feb;41(1):82-93. doi: 10.1080/00224490409552216. PMID 15216427
- [Background] Wierman ME, Nappi RE, Avis N, Davis SR, Labrie F, Rosner W, Shifren JL. Endocrine aspects of women's sexual function. J Sex Med. 2010 Jan;7(1 Pt 2):561-85. doi: 10.1111/j.1743-6109.2009.01629.x. PMID 20092453
- [Result] Scavello I, Maseroli E, Di Stasi V, Cipriani S, Verde N, Magini A, Maggi M, Vignozzi L. Nomegestrol acetate/17beta-estradiol does not negatively alter the vascular resistance of clitoral arteries: a prospective, exploratory study. Int J Impot Res. 2020 Mar;32(2):239-247. doi: 10.1038/s41443-019-0162-7. Epub 2019 Jul 1. PMID 31263248